CLINICAL TRIAL: NCT02524288
Title: A Phase 3, Single Arm, Clinical Trial to Study the Contraceptive Efficacy and Safety of the MK-8342B (Etonogestrel + 17β-Estradiol) Vaginal Ring in Healthy Women 18 Years of Age and Older, At Risk for Pregnancy
Brief Title: Efficacy and Safety of Etonogestrel + 17β-Estradiol Vaginal Ring in Women at Risk for Pregnancy (MK-8342B-061)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated by the Sponsor due to a business decision to discontinue product development for reasons unrelated to safety or efficacy outcomes.
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8342B-061
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — Contraceptive Devices, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ENG-E2 125 μg/300 μg (Experimental): Participants will receive up to 13 cycles of ENG-E2 125 μg/300 μg. Each cycle will consist of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: ENG-E2 125 μg/300 μg vaginal ring

INTERVENTIONS:
Drug: ENG-E2 125 μg/300 μg vaginal ring — Up to 13 cycles of ENG-E2 125 μg/300 μg administered intravaginally, each cycle consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.

SUMMARY:
The purpose of this study is to assess the contraceptive efficacy of the Etonogestrel (ENG) + 17β-Estradiol (E2) vaginal ring in women between 18 and 35 years of age based on the number of in-treatment pregnancies as expressed by the Pearl Index (PI). The study will also assess the safety and tolerability of the ENG-E2 vaginal ring.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female at risk for pregnancy and seeking contraception.
* Willing to use a hormonal contraceptive vaginal ring for up to 13 treatment cycles, and not intending to use any other form of contraception.
* Body mass index (BMI) of ≥18 and <38 kg/m2.
* Willing to adhere to use of vaginal ring and all required trial procedures.

Exclusion Criteria:

* Cardiovascular risks and disorders, including history of venous thromboembolic [VTE] events, arterial thrombotic or thromboembolic [ATE] events, transient ischemic attack, angina pectoris, or claudication; at higher risk of VTE events due to recent prolonged immobilization, plans for surgery requiring prolonged immobilization, or a hereditary or acquired predisposition or elevated risk for venous or arterial thrombosis; currently smoking or uses tobacco/nicotine containing products and is ≥35 years of age; uncontrolled or severe hypertension; history of severe dyslipoproteinemia; <35 years of age with a history of migraine with aura or focal neurological symptoms or ≥35 years of age with a history of migraines with or without aura or focal neurologic symptoms; diabetes mellitus with end-organ involvement or >20 years duration; multiple cardiovascular risk factors such as older age, obesity, inadequately controlled hypertension, use of tobacco/ nicotine products, or inadequately controlled diabetes.
* Gastrointestinal disorders, including history of pancreatitis associated with severe hypertriglyceridemia; clinically significant liver disease, including active viral hepatitis or cirrhosis.
* Other medical disorders, including history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer; any disease that may worsen under hormonal treatment such as disturbances in bile flow, systemic lupus erythematosus, pemphigoid gestationis or idiopathic icterus during previous pregnancy, middle-ear deafness, Sydenham chorea, or porphyria; known allergy/sensitivity or contraindication to investigational product or its excipients; history of drug or alcohol abuse or dependence.
* Recent, current, or suspected pregnancy; or has not had at least 2 menstrual cycles or has not completed two 28-day cycles of a hormonal contraceptive (pill, patch or ring) following a recent pregnancy; or is breastfeeding.
* Gynecologic conditions: has gonorrhea, chlamydia, or trichomonas or symptomatic vaginitis/cervicitis; has abnormal cervical Pap test or positive high-risk human papillomavirus (HPV) test at screening or documented within 3 years of screening; currently using an intrauterine device/ intrauterine system (IUD/ IUS) or contraceptive implant; within past 6 months has had undiagnosed (unexplained) abnormal vaginal bleeding or any abnormal bleeding expected to recur during trial; has stage 4 pelvic organ prolapse (1 cm beyond introitus) or lesser degrees of prolapse with history of difficulty retaining tampons, vaginal rings, or other products within vagina.
* Has used investigational drug and/or participated in other clinical trial within past 8 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1941 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ENG-E2 125 μg/300 μg: Participants were to receive up to 13 cycles of Etonogestrel (ENG) 125 μg and 17β-Estradiol (E2) 300 μg. Each cycle would consist of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
Period: Overall Study
Arm/Group | ENG-E2 125 μg/300 μg
Started | 1941
Treated | 1936
Completed | 0
Not Completed | 1941
Not completed — Adverse Event | 115
Not completed — Lost to Follow-up | 216
Not completed — Non-Compliance With Protocol | 32
Not completed — Non-Compliance With Study Drug | 14
Not completed — Pregnancy Wish | 6
Not completed — Protocol Violation | 6
Not completed — Screen Failure | 2
Not completed — Site Discontinued Study Participation | 1
Not completed — Study Terminated By Sponsor | 1417
Not completed — Subject Moved | 32
Not completed — Withdrawal by Subject | 76
Not completed — Pregnancy | 22
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | ENG-E2 125 μg/300 μg
Number analyzed (Participants) | 1941
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1941
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of In-Treatment Pregnancies Per 100 Woman-Years of Exposure in Participants 18-35 Years of Age (Pearl Index)
Description: The Pearl Index is the number of in-treatment pregnancies with a conception date in any of the in-treatment cycles, divided by all treatment cycles in each participant from the first treatment cycle to the last treatment cycle (due either to discontinuation or completion), regardless of whether a treatment cycle was "at risk" or not. One woman-year is defined as 13 treatment cycles x 28 days. These efficacy results should be interpreted with caution. Due to the discontinuation of product development and early trial termination, the number of "at risk" treatment cycles in the denominator is based on uncleaned diary data.
Time Frame: Up to 1 year (13 28-day cycles)
Population: All participants assigned to treatment who inserted at least 1 ENG-E2 ring, and who had at least 1 "at risk" treatment cycle, or participants with a treatment cycle (at risk or not) in which a pregnancy had occurred (i.e., treatment cycle containing an estimated conception date for a pregnancy).
Measure: Number; unit: Pregnancies per 100 woman years
Arm/Group | ENG-E2 125 μg/300 μg
Number analyzed (Participants) | 1574
Pregnancies per 100 woman years | 4.32

2. Primary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: From insertion of the first vaginal ring up to and including 14 days after removal of the last vaginal ring (up to approximately 1 year)
Population: All randomized participants in whom at least 1 vaginal ring was inserted.
Measure: Number; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg
Number analyzed (Participants) | 1936
Participants | 830

3. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All randomized participants in whom at least 1 vaginal ring was inserted.
Measure: Number; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg
Number analyzed (Participants) | 1936
Participants | 112

4. Primary Outcome: Number of Participants With One or More Drug-related AEs
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the Sponsor's product, is also an AE. An investigator who is a qualified physician determined whether an AE is drug-related.
Time Frame: as for outcome 2
Population: All randomized participants in whom at least 1 vaginal ring was inserted.
Measure: Number; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg
Number analyzed (Participants) | 1936
Participants | 439

5. Primary Outcome: Number of Participants Who Discontinued Treatment Due to a Drug-related AE
Description: as for outcome 4
Time Frame: as for outcome 2
Population: All randomized participants in whom at least 1 vaginal ring was inserted.
Measure: Number; unit: Participants
Arm/Group | ENG-E2 125 μg/300 μg
Number analyzed (Participants) | 1936
Participants | 91

ADVERSE EVENTS:
Time Frame: From insertion of the first vaginal ring up to and including 14 days after removal of the last vaginal ring (up to approximately 1 year)
Description: All randomized participants in whom at least 1 vaginal ring was inserted.
Arm/Group | ENG-E2 125 μg/300 μg
Serious Adverse Events (participants affected / at risk) | 12/1936
Other Adverse Events (participants affected / at risk) | 0/1936
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENG-E2 125 μg/300 μg (N=1936)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Results for the Pearl Index should be interpreted with caution. Due to the discontinuation of product development and early trial termination, the number of "at risk" treatment cycles in the denominator is based on uncleaned diary data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.